CLINICAL TRIAL: NCT04756284
Title: A Pilot Study to Evaluate the PhageTech Virus BioResistor inDetecting Combinations of Bladder Cancer Biomarkers inPatients Under Active BCa Surveillance
Brief Title: Evaluation of the PhageTech Virus BioResistor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PhageTech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VBRm BCA-01
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bladder Tumor Positive: Patients with previous bladder cancer diagnosis; any stage and histological type, undergoing cystoscopy or suspected bladder tumor undergoing surveillance cystoscopy.
- Bladder Tumor Negative: Patients with no suspected bladder tumor.

SUMMARY:
To evaluate the effectiveness of the PhageTech Virus BioResistor to detect bladder cancer biomarkers.

DETAILED DESCRIPTION:
This study will sample urine provided by bladder cancer patients as part of their normal routine surveillance screening. No additional effort will be required from the patients and only modest additional effort from the study staff. Some de-identified patient medical information may also be requested, including concominant medications, relevant current or previous diseases, prior bladder cancer interventions and other relevant information to ensure there are no interfering substances or other confounders that could affect study results. There is no risk to patients as the normal diagnostics for bladder cancer will be followed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 18 years
2. Previous bladder cancer diagnosis; any stage and histological type, undergoing cystoscopy
3. Patients with suspected bladder tumor undergoing surveillance cystoscopy
4. Patients must provide written Informed Consent.

Exclusion Criteria:

1. Patients unable or unwilling to sign the informed consent
2. Age < 18 years
3. Known HIV/HCV/HBV (information from clinical history).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will sample urine provided by bladder cancer patients as part of their normal routine surveillance screening. No additional effort or samples will be required from the patients. Results from this study will not be used for any of the normal physician diagnostic process. Patients will have a suspected bladder tumor undergoing cystoscopy or a history of bladder cancer undergoing surveillance cystoscopy. Patients who have had a positive diagnosis of bladder cancer, but have not yet had a tumor resection (known BCa positive patients) are highly desirable for this study. It is anticipated that the majority of samples collected will be negative. In the case of a known BCa positive patient, the sponsor is requested
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-08 (Estimated); Primary Completion 2021-11-11 (Estimated); Study Completion 2021-11-11 (Estimated)

PRIMARY OUTCOMES:
Successful identification of bladder tumor biomarkersBiomarkers in Patients Under Active BCa Surveillance | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Saint John's Health Center and the Saint John's Cancer Institute, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided